CLINICAL TRIAL: NCT00604682
Title: Open-Label, Single-Arm Pilot Study to Evaluate the Pharmacodynamics, Pharmacokinetics, Safety, and Preliminary Efficacy of CC10004 in Subjects With Severe Plaque Type Psoriasis
Brief Title: Open-Label,Single-Arm Pilot Study to Evaluate the Pharmacodynamics, Pharmacokinetics, Safety, and Preliminary Efficacy of CC1004 in Subjects With Severe Plaque Type Psoriasis
Acronym: PSOR-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-001
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Administration of CC10004 (Experimental)
  Interventions: Drug: CC10004

INTERVENTIONS:
Drug: CC10004 — 2 X 10 mg caps taken once daily for a daily dose of 20 mg. Must be taken upon awakening and fasted
  Other Names: Apremilast

SUMMARY:
Open label study for patients with severe plaque type psoriasis. This study is looking to evaluate the pharmacodynamic effect of CC10004 when taken for 29 days in reducing the epidermal thickness in subjects with severe placque type psoriasis.

ELIGIBILITY:
Inclusion Criteria

* Must understand and voluntarily sign an informed consent form
* Must be age > or = to 18 years to 65 years at the time of singing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must have a history of severe plaque type psoriasis for at least 6 months, and at least a 15% affected total body surface area (BSA)
* Must meet the following clinical laboratory criteria:
* White Blood Cell Count > or = to 3000/cu mm and < 20,000/cu mm
* Platelet count > or = to 100,000/microliters
* Serum creatinine < or = to 1.5 mg/dl
* Total bilirubin < or = to 2.0 mg/dl
* AST (SGOT) and ALT (SGPT) < or = to 1.5 X ULN
* Must have a psoriatic plaque > or = to 2.5 cm in diameter (for biopsy)
* Must be candidate for photo/systemic therapy (a subject is considered a candidate for photo/systemic therapy if a clinician judges that the subject requires any systemic therapy (e.g., ultraviolet light B(UVB), Psoralens and long-wave ultraviolet radiation (PUVA), cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, tacrolimus, azathioprine)to control psoriasis whether or not that subject has a history of receiving systemic therapy)
* Women of child bearing potential (WCBP) must have a negative urine pregnancy test at Screening (Visit 1). In addition, sexually active WCBP must agree to use two forms of adequate forms on contraception throughout the trial.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality , or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Current erythrodermic, guttate, or pustular psoriasis
* Use of medication that is metabolized by the CYP3A4 or CYP2A6 pathways within the 14 days of study medication initiation and/or required use of such medication during study treatment.
* Drinking or ingesting grapefruits, grapefruit juice or grapefruit containing products within 14 days of study medication initiation
* Use of topical therapy ( topical steroids, topical vitamin A or D analog preparations, tacrolimus, pimecrolimus, or anthralin) within 14 days of study medications initiation (Exception: Non-medicated emollients and tar shampoo will be allowed)
* Use of systemic therapy for psoriasis
* Use or phototherapy within 28 days of study medication initiation
* Use Humira or Remicade within 3 months of study medication initiation
* Use of Enbrel within 56 days of study medication initiation
* Use of Raptiva within 56 days of study medication initiation
* Use of Amevive within 6 months of study medication initiation
* Use of any investigational drug within 30 days of study medication initiation or 5 half lives if known
* History of clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic insufficiency disease or other major diseases
* Clinically significant abnormality on 12-lead ECG at screening
* Positive HIV, Hepatitis B or Hepatitis C laboratory result at screening
* History of active tuberculosis within previous 3 years
* Clinically significant abnormality on the chest x-ray at screening or on CXR taken within 6 months of screening
* History of positive purified protein derivative (PPD) test at screening
* History of malignancy within previous five years
* Evidence of skin conditions at the time of screening visit other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2005-10-01 (Actual); Study Completion 2005-12-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacodynamic effect of orally administered CC10004 when taken for 29 days in reducing epidermal thickness in subjects with severe plaque-type psoriasis. | 29 days

SECONDARY OUTCOMES:
To evaluate the safety of orally administered CC10004 in subjects with severe plaque-type psoriasis during the treatment and follow up phases. | 58 days
To explore the clinical efficacy of orally administered CC10004 when taken for 29 days in subjects with severe plaque-type psoriasis. | 29 days
To explore the clinical efficacy of CC10004 when taken for 29 days in subjects with psoriatic arthritis. | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine, New York, New York
  - Mt Sinai School of Medicine, New York, New York

REFERENCES:
- [Background] Gottlieb AB, Strober B, Krueger JG, Rohane P, Zeldis JB, Hu CC, Kipnis C. An open-label, single-arm pilot study in patients with severe plaque-type psoriasis treated with an oral anti-inflammatory agent, apremilast. Curr Med Res Opin. 2008 May;24(5):1529-38. doi: 10.1185/030079908x301866. Epub 2008 Apr 16. PMID 18419879